CLINICAL TRIAL: NCT05521243
Title: An Exploratory Investigation of a Supplement to Enhance Sleep Quality and Quantity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beam (Industry)
Collaborators: Citruslabs (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Other
Other Study IDs: 20241
Record Dates: First submitted 2022-08-24; First posted 2022-08-30 (Actual); Last update posted 2022-11-08 (Actual); Status verified 2022-11

CONDITIONS: Sleep; Sleep Disturbance; Sleep Hygiene
Keywords: Sleep; Sleep Disturbance; Sleep Quality; Sleep Quantity
MeSH Terms: conditions — Parasomnias; Sleep Hygiene; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo + Dream Powder (Experimental): Participants take the placebo product for two weeks, followed by the Dream Powder intervention product for four weeks.
  Interventions: Dietary Supplement: Beam Organics Dream Powder; Dietary Supplement: Placebo
- Placebo + Dream Powder Extra Strength (Experimental): Participants take the placebo product for two weeks, followed by the Dream Powder Extra Strength intervention product for four weeks.
  Interventions: Dietary Supplement: Beam Organics Dream Powder Extra Strength; Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Beam Organics Dream Powder — The Dream Powder and Dream Powder Extra Strength both use nano hemp, reishi, magnesium. L-theanine, and melatonin to promote a healthy sleep pattern
  Arms: Placebo + Dream Powder
Dietary Supplement: Beam Organics Dream Powder Extra Strength — The Dream Powder and Dream Powder Extra Strength both use nano hemp, reishi, magnesium. L-theanine, and melatonin to promote a healthy sleep pattern
  Arms: Placebo + Dream Powder Extra Strength
Dietary Supplement: Placebo — The main ingredients in the placebo are:
  Coconut milk powder, cocoa, cinnamon, monk fruit, natural vanilla flavor

SUMMARY:
This double-blind study will examine the effectiveness of Dream Powder and Dream Powder Extra Strength over a six week period. The main outcomes of interest will be sleep quantity and quality, as well as self-reported changes in sleep across the study period.

ELIGIBILITY:
Inclusion Criteria:

* Self-reported issues with sleep Must be in good overall health with no unstable medical conditions Must own a wearable sleep tracker (i.e., Apple Watch, "FitBit", "Whoop", etc.) Must be willing to discontinue any supplements meant to assist with sleep.

Exclusion Criteria:

* Females who are pregnant or breastfeeding Diagnosis of insomnia or sleep apnea Taking a prescription medication that affects sleep Anyone with a pre-existing condition that would prevent them from adhering to the protocol Anyone with a known history of past severe allergic reactions

Ages: 24 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2022-05-09 (Actual); Primary Completion 2022-09-30 (Actual); Study Completion 2022-09-30 (Actual)

PRIMARY OUTCOMES:
Perceived Changes in Sleep Quality as reported by questionnaires | 6 Weeks
  Examined across the six week trial with questionnaires. These questionnaires will occur at Baseline, Week 2, Week 4, and Week 6, and will gather information about their ability to fall asleep, stay asleep, and the overall amount of sleep they get on average during the past week.
Perceived Changes in Sleep Quantity as reported by questionnaires | 6 weeks
  Examined across the six week trial with questionnaires. These questionnaires will occur at Baseline, Week 2, Week 4, and Week 6, and will gather information about their ability to fall asleep, stay asleep, and the overall amount of sleep they get on average during the past week.
Perceived Changes in Sleep Habits as reported by Questionnaires | 6 weeks
  Examined across the six week trial with questionnaires. These questionnaires will occur at Baseline, Week 2, Week 4, and Week 6, and will gather information about their ability to fall asleep, stay asleep, and the overall amount of sleep they get on average during the past week.
Participant Perceptions of Sleep | 6 weeks
  Examined across the six week trial with questionnaires. These questionnaires will occur at Baseline, Week 2, Week 4, and Week 6, and will gather information about their ability to fall asleep, stay asleep, and the overall amount of sleep they get on average during the past week.

SECONDARY OUTCOMES:
Examine changes in device measured sleep across the six week trial. | 6 Weeks
  Sleep will be measured with fitness trackers to provide an objective outcome measure of sleep across the six week trial. Both sleep time and sleep quality will be examined. Participants will report their sleep data from the previous week at Baseline, Week 2, Week 4, and Week 6.

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Hill, PhD, Principal Investigator — Citruslabs
Locations (1):
- Citruslabs, Santa Monica, California, United States

IPD SHARING:
Plan to Share IPD: Undecided